CLINICAL TRIAL: NCT05215964
Title: The Association Between Skeletal Muscle Mass and Severity of Polycystic Liver Disease and Polycystic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006139RINA
Record Dates: First submitted 2021-05-28; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-10

CONDITIONS: Polycystic Kidney Diseases; Polycystic Liver Disease; Muscle Loss
MeSH Terms: conditions — Polycystic Kidney Diseases; Polycystic liver disease; Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — hemogram, complete blood count, CBC renal function: BUN, Cr electrolytes: Na, K, Ca, P hypertension: plasma renin activity, aldosterone inflammation: CRP, IL-6、TNF-α、IL-1 liver function: AST, ALT, Albumin, T-Bil, PT, INR muscle: CPK, myostatin adipose: Cholesterol, TG, HDL, LDL, adiponectin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAE arm: Patients will receive TAE
  Interventions: Procedure: Renal artery embolization

INTERVENTIONS:
Procedure: Renal artery embolization — After catheterization of renal arteries, multiple coils are applied to embolize renal arteries until blood flow stasis

SUMMARY:
Primary sarcopenia is used to describe aging and progressed with the physiologic decline. Secondary sarcopenia is associated many chronic disease, including acquired immune deficiency syndrome, cancer, chronic heart failure, chronic lung disease, liver cirrhosis, chronic kidney disease and rheumatoid arthritis. In the past, nutrition status is evaluated by body mass index, mid-upper -arm circumference and serum albumin. Bioelectrical impedance analysis is also a common method to measured body composition, but bioelectrical impedance analysis will be affected by tissue edema and ascites. In contrast, cross-section imaging, such as computed tomography and magnetic resonance can analyzed abdominal muscle and fat accurately.

Since computed tomography and magnetic resonance imaging can evaluate the severity of polycystic liver and kidney disease. Investigators can use cross section imaging at 3rd lumber level to separate skeletal muscle and fat tissue. Previous studies showed the quantity and quality of abdominal muscle are important prognostic factor after liver transplantation. Besides, chronic kidney disease and receiving renal placement therapy lead protein catabolism and make patients with end stage renal disease have sarcopenia. Finally, patients with polycystic liver and kidney disease have organomegaly, which causes abdominal distention and poor appetite. Therefore, the aim of this study is to observe the association between skeletal muscle mass and the severity of disease and to study whether change in hepatic and renal volumes is associated with change in muscle mass.

DETAILED DESCRIPTION:
The imaging study (CT or MRI) will be performed within one month before the procedure to measure total kidney volume and psoas muscle area.

The procedure will use transcatheter embolization to renal artery. The follow-up imaging study will be performed six months after the procedure to measure total kidney volume and psoas muscle area..

ELIGIBILITY:
Inclusion Criteria:

* Polycystic related disease with medical images (CT or MRI) diagnosed
* Aged over 20 years

Exclusion Criteria:

* Lack of Bio-exam or medical images
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Retrospective group：participants had done TAE procedures since from January 2015 to July 2020.
  2. Prospective group：two groups, 1. willing to receive cysts control procedures, 2. medical images follow up only
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Total psoas muscle change | 6 months by imaging study
  The change of psoas muscle area before and after procedures.

SECONDARY OUTCOMES:
Total kidney volume change | 6 months by imaging study
  The change of total kidney volume before and after procedures

CONTACTS AND LOCATIONS:
Overall Officials: Ared Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided